CLINICAL TRIAL: NCT07367360
Title: A Comparative Analysis of Stretching Exercise and Pregnancy Exercise on Sleep Quality in Pregnancy: A Quasi Experiment
Acronym: CESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Polytechnic of Palangka Raya (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 121/II/KE.PE/2024; 121/II/KE.PE/2024 (Other Grant/Funding Number: Health Polytechnic of Palangka Raya)
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sleep Deprivation; Sleep Wake Disorders; Pregnancy; Anxiety Disorders; Stretching Exercises; Relaxation Therapy
Keywords: Pregnancy; Sleep Deprivation; Anxiety; Stretching Exercises; Exercise Therapy
MeSH Terms: conditions — Sleep Deprivation; Sleep Wake Disorders; Anxiety Disorders | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with each group receiving a distinct exercise intervention. Clinics use their own staff and routines, creating natural variation in session delivery.
  Both groups follow structured exercise programs for pregnant women in the third trimester:
  Intervention Group: Traditional pregnancy exercises per Indonesian Ministry of Health guidelines.
  Control Group: Stretching focused on flexibility and relaxation. Participants complete two supervised sessions weekly for three weeks (45-60 minutes/session) and receive home practice materials. Sleep quality, anxiety, physical activity, and health indicators are measured before and after to compare changes. The design enables researchers to assess the impact of two exercise approaches on sleep quality, accounting for individual differences.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm take part in a structured traditional pregnancy exercise program designed specifically for women in the third trimester. The program follows guidelines from the Indonesian Ministry of Health and includes gentle movements, breathing techniques, posture training, pelvic floor exercises, and relaxation components intended to support comfort and well-being during late pregnancy. Sessions are conducted twice per week for three weeks, with each session lasting approximately 45-60 minutes and led by trained midwives or instructors at the participating clinic. Participants also receive printed and video materials to support safe practice at home. The intervention aims to improve sleep quality, reduce physical discomfort, and promote relaxation.
  Interventions: Other: Traditional Pregnancy Exercise Group; Other: Stretching Exercise Group (Control)
- Control group (Experimental): Participants in the control group take part in a stretching exercise program designed to promote flexibility, reduce muscle tension, and support overall comfort during late pregnancy. The program consists of gentle, low-intensity stretching movements that target major muscle groups commonly affected during the third trimester, such as the back, hips, legs, and shoulders. Sessions are conducted twice per week for three weeks, with each session lasting approximately 45-60 minutes and guided by trained clinic staff. The stretching routine is simple, safe, and suitable for pregnant women, and participants receive printed and video materials to help them practise at home. This intervention serves as a comparison condition to evaluate whether traditional pregnancy exercise offers additional benefits for sleep quality and anxiety beyond those provided by basic stretching.
  Interventions: Other: Traditional Pregnancy Exercise Group; Other: Stretching Exercise Group (Control)

INTERVENTIONS:
Other: Traditional Pregnancy Exercise Group — A structured exercise program for third-trimester pregnant women, following the Indonesian Ministry of Health guidelines. Includes breathing techniques, gentle movements, posture training, pelvic floor exercises, and relaxation. Conducted twice weekly for 3 weeks, 45-60 minutes per session, led by trained clinic staff.
  Other Names: Traditional Pregnancy Exercise
Other: Stretching Exercise Group (Control) — A low-intensity stretching routine targeting major muscle groups to reduce tension and support comfort during late pregnancy. Conducted twice weekly for 3 weeks, 45-60 minutes per session, guided by trained clinic staff.
  Other Names: Stretching Exercise

SUMMARY:
The goal of this clinical trial is to learn whether pregnancy exercise or stretching exercise can improve sleep quality in third trimester pregnant women who experience sleep disturbances. The main questions it aims to answer are:

* Does traditional pregnancy exercise improve sleep quality more effectively than stretching exercise?
* Does either type of exercise reduce anxiety levels that may affect sleep? Researchers will compare a pregnancy exercise group with a stretching exercise group to see whether one approach leads to better sleep quality.

Participants will:

* Attend guided exercise sessions twice a week for three weeks
* Complete questionnaires about sleep quality, anxiety, and physical activity
* Have basic health measurements taken (blood pressure, weight, height) before and after the program

This study hopes to show whether moderate exercise can help pregnant women sleep better during the third trimester.

DETAILED DESCRIPTION:
Sleep problems are very common during pregnancy, especially in the third trimester, when physical discomfort, hormonal changes, and anxiety often make it difficult for women to rest well. Poor sleep can affect a mother's physical and emotional health, contribute to stress and fatigue, and may even influence labour and delivery outcomes. Although exercise is widely recommended during pregnancy, there is still limited research on which types of exercise are most helpful for improving sleep.

This study aims to better understand whether traditional pregnancy exercise or stretching exercise can help improve sleep quality among third trimester pregnant women living in Palangka Raya, Central Kalimantan. Both types of exercise are commonly used in Indonesia, but their specific effects on sleep have not been directly compared in a structured research setting.

A total of 60 pregnant women between 28 and 30 weeks of gestation will take part in the study. Participants are divided into two groups based on the midwifery clinic where they receive care. One group will participate in traditional pregnancy exercise, a structured program developed by the Indonesian Ministry of Health that includes breathing techniques, gentle movements, and relaxation. The other group will take part in a stretching exercise program, which focuses on improving flexibility and reducing muscle tension.

Both programs run for three weeks, with two supervised sessions per week, each lasting about 45-60 minutes. Participants also receive a booklet and video materials so they can practise at home.

To understand how these exercises affect sleep, participants complete several assessments before and after the program:

* Pittsburgh Sleep Quality Index (PSQI) to measure sleep quality
* Hamilton Anxiety Rating Scale (HARS) to assess anxiety levels
* International Physical Activity Questionnaire (IPAQ) to evaluate overall physical activity
* Basic health measurements such as blood pressure, weight, and height

By comparing the results from both groups, the study will explore whether one type of exercise leads to greater improvements in sleep quality or anxiety. The findings may help midwives, health workers, and pregnant women choose effective, safe, and accessible exercise options to support better sleep during late pregnancy.

The goal of this research is to promote healthier pregnancies by finding easy, non-medicinal ways to help expectant mothers sleep better and enhance their overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester (28-30 weeks of gestation at enrollment).
* Having sleeping disturbance complaints.
* Aged more than 19 years old.
* Being under prenatal clinical follow-up
* Not having or participating in specific treatment for sleeping disturbance in the last 3 months
* Able to participate in light to moderate physical activity as assessed by clinic staff.
* Signing informed consent for study participation.

Exclusion Criteria:

* Failure to attend at least 70% of the 12 planned sessions
* Having pregnancy complication.
* Gestational ages < 28 or > 30 weeks.
* Not having bleeding history, abortion.
* Not having multiple pregnancy.
* Medical or obstetric conditions that make exercise unsafe (e.g., preeclampsia, placenta previa, risk of preterm labor, uncontrolled hypertension)
* Current participation in another structured exercise program.
* Severe musculoskeletal problems that limit movement.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is open only to women who are currently pregnant. Because the research focuses on sleep quality and exercise during the third trimester of pregnancy, only individuals who identify as female and are carrying a pregnancy can take part. People who are not pregnant or who are not biologically able to become pregnant are not eligible for this study.
Enrollment: 60 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI), measured at baseline and after the 3-week intervention period | From enrollment and baseline measurement to completion of the 3-week exercise program
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated questionnaire that evaluates sleep patterns over the previous one-month period. The PSQI consists of 19 self-rated items** that generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 to 3, and the scores are summed to produce a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality. A global PSQI score greater than 5 is commonly used to define poor sleep quality. Participants complete the PSQI at baseline and again after the three-week intervention period to determine changes in sleep quality associated with the exercise programs.

CONTACTS AND LOCATIONS:
Overall Officials: Vissia Didin Ardiyani, Dr, Study Chair — Health Polytechnic of Palangka Raya
Locations (1):
- Midwifery clinics, Palangkaraya, Central Kalimantan, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive health information from pregnant women, and sharing it could compromise participant privacy and confidentiality. Additionally, the study was not designed with data-sharing agreements or infrastructure in place to support secure external access.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT07367360/Prot_SAP_ICF_000.pdf